CLINICAL TRIAL: NCT06666283
Title: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AP303 Following 2-week Oral Administration in Diabetic Kidney Disease Patients With Renal Impairment.
Brief Title: A Study to Evaluate the Safety, Tolerability, PK and PD of AP303 in DKD Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alebund Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP303-PK-03
Record Dates: First submitted 2024-10-18; First posted 2024-10-30 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AP303 (Experimental)
  Interventions: Drug: AP303 150μg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo 150μg

INTERVENTIONS:
Drug: AP303 150μg — AP303 Tablet 150μg QD
  Arms: AP303
Drug: Placebo 150μg — Placebo Tablet 150μg QD
  Arms: Placebo

SUMMARY:
The study will be a single center, double-blind, randomized, placebo-controlled study to evaluate the safety, tolerability, PK and PD of AP303 following 2-week oral administration to Diabetic Kidney Disease patients.

DETAILED DESCRIPTION:
Eligible patients will be enrolled into one of the two dose cohorts, each cohort will include 9 participants randomized to AP303 and placebo at a 2:1 ratio (6 on AP303 and 3 on placebo).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants, ≥30 years of age at the time of signing the informed consent form.
2. BMI (body mass index) 18-30 kg/m².
3. Patient has a clinical diagnosis of Type 2 Diabetes Mellitus and is taking at least one type of hypoglycemic drugs, before screening visits, the doses of hypoglycemic drugs, including insulin, need to be stable for at least two weeks..
4. Patient must be on a stable dose of angiotensin converting anzyme inhibitior (ACEI) or Angiotensin II receptor blockers (ARB) for at least 4 weeks prior to screening.
5. Hemoglobin A1c ≥6.5% but ≤10.5% at the screening visit.
6. Estimated GFR ≥30 mL/min/1.73m² but < 60 mL/min/1.73m² at the screening visit.
7. Urinary albumin to creatinine ratio ≥ 30 mg/g at the screening visit.

Exclusion Criteria:

1. Chronic kidney disease other than type 2 diabetic kidney disease.
2. Patient receiving corticosteroid immunotherapy or other immunosuppressants (such as calcineurin inhibitors ciclosporin, cyclophosphamide, or mycophenolate mofetil) in the past 3 months before screening.
3. Recently having acute kidney injury or received renal surgery within the last 6 months before screening visit, or have received renal transplantation.
4. Congestive heart failure classified New York Heart Association (NYHA) class II to IV within the last 3 months before the screening visit.
5. Peripheral edema above the ankle level at the screening or randomization visit.
6. Confirmed (based on the average of 2 separate resting blood pressure measurements in a sitting position, after at least 5 minutes rest) systolic BP greater than 160 or less than 90 mmHg, and diastolic BP greater than 100 or less than 50 mmHg at screening.
7. Myocardial infarction, acute coronary syndrome, stroke or transient ischemic attack, cardiovascular surgery within 6 months prior to the screening visit.
8. Abnormalities of ECG parameters and abnormal shape of ECG wave on screening ECG: e.g.

   * QTc interval (QTcF > 450 ms for male and QTcF > 470 ms for female) based on the average interval on triplicate ECGs obtained after 5 minute's rest in a supine position
   * Notable resting bradycardia (mean HR < 40 bpm)
   * Notable resting tachycardia (mean HR > 100 bpm)
   * ECG with QRS and/or T wave judged to be unfavorable for a consistently accurate QT measurement (e.g., neuromuscular artifact that cannot be readily eliminated, indistinct QRS onset, low amplitude T wave, merged T- and U-waves, prominent U waves)
   * Any other significant abnormality
9. Implantation of cardiac pacemaker or clinically significant arrhythmia, e.g. atrial fibrillation, atrial flutter, right or left bundle branch block, Wolf-Parkinson-White Syndrome.
10. Current or previous treatment with a thiazolidinedione (e.g., medications containing pioglitazone or rosiglitazone, like Actos, Avandia, ActoplusMet, Avandamet, Avandaryl), PPARa agonist (like fenofibrate) or any dual/multiple PPARa/g agonist (e.g., Chiglitazar Sodium) in the 3 months preceding screening visit.
11. Previous treatment with CYP2C8 inducer or strong/moderate inhibitor (refer to the list in Appendix 4) in the 1 month preceding screening visit.
12. Chronic therapy with non-steroidal anti-inflammatory drugs (NSAIDs) (except prophylactic stable low dose aspirin, defined as its dose not higher than 100 mg daily; paracetamol/acetaminophen was allowed) in the last month before screening.
13. ALT or AST >1.5 × ULN, or laboratory tests revealed other clinically significant abnormalities in liver function at screening.
14. Creatine phosphokinase (CPK) elevated > 3 x ULN at screening visit or history of drug-induced myopathy.
15. History of malignancy within 5 years before screening (exceptions: squamous and basal cell carcinomas of the skin and carcinoma of the cervix in situ, or a malignancy that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence).
16. Participants who have had significant acute infection, e.g., COVID-19, influenza, local infection, acute gastrointestinal symptoms or any other clinically significant illness within two weeks before study drug administration.
17. Positive test at screening of any of the following: Hepatitis B (HBsAg), Hepatitis C (HCVAb), human immunodeficiency virus (HIV Ab) or syphilis AB.
18. Dosed with a small-molecule investigational drug within 3 months, or biologic investigational drug within 3 months or 5 half-lives (whichever is the longer) prior to first dose of this study.
19. History of drug and/or alcohol abuse or addiction. History (within 3 months of screening) of alcohol consumption exceeding 3 and 2 standard drinks per day on average (1 standard drink = 10 grams of alcohol) for male and female, respectively.
20. Within 2 weeks prior to admission, use of >5 cigarettes or equivalent nicotine-containing product per day.
21. Medical or social conditions that would potentially interfere with the participant's ability to comply with the study visit schedule or the study assessments.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
Cmax | Day 1, Day 14
  Maximum observed plasma concentration
Tmax | Day 1, Day 14
  Time to maximum observed plasma concentration
AUC0-24h | Day 1
  Area under the plasma concentration versus time curve up to 24 hours
AUC0-last | Day 1
  Area under the plasma concentration versus time curve up to the last measurable concentration
AUC0-inf | Day 1
  Area under the plasma concentration versus time curve extrapolated to infinity
AUC0-t | Day 14
  Area under the plasma concentration-time curve for a dosing interval
t1/2 | Day 1, Day 14
  Apparent terminal half-life, computed as ln(2)/λz
CL/F | Day 1
  Apparent oral clearance calculated from Dose/ AUC0-inf
V/F | Day 1, Day 14
  Apparent volume of distribution of oral drug
Cav | Day 14
  Average plasma concentration
Ctrough | Day 3-14
  Trough plasma concentration
Rac | Day 3-14
  Ratio of accumulation
Incidence and severity of adverse events | Day 1-28
  Incidence and severity of adverse events
Incidence of laboratory abnormalities, based on hematology, clinical chemistry, coagulation and urinalysis test results | Day 1-28
  Incidence of laboratory abnormalities, based on hematology, clinical chemistry, coagulation and urinalysis test results
Effect of AP303 on ECG parameters | Day 1-28
  Change of Heart rate in beats/min
Effect of AP303 on ECG parameters | Day 1-28
  change of QT in ms
Effect of AP303 on ECG parameters | Day 1-28
  Change of PR in ms
Effect of AP303 on ECG parameters | Day 1-28
  Change of QRS in ms
Effect of AP303 on ECG parameters | Day 1-28
  Change of QTcF in ms
Effect of AP303 on ECG parameters | Day 1-28
  Change of QTcB in ms
Vital signs（Systolic blood pressure） | Day 1-28
  Change of systolic blood pressure
Effect of AP303 on physical examination result | Day 1-28
  Number of pariticipants with abnormal physical examination findings by nature and severity
Body weight | Day 1-28
  Change of body weight
Vital signs (Diastolic blood pressure) | Day1-28
  Change of diastolic blood pressure
Vitlal signs (Body temperature) | Day 1-28
  Change of body temperature
Effect of AP303 on ECG parameters | Day 1-28
  Number of participants with abnormal QTcB.
Effect of AP303 on ECG parameters | Day 1-28
  Number of participants with abnormal QTcF
Effect of AP303 on ECG parameters | Day 1-28
  Number of participants with abnormal QRS
Effect of AP303 on ECG parameters | Day 1-28
  Number of participants with abnormal PR
Effect of AP303 on ECG parameters | Day 1-28
  Number of participants with abnormal QT
Effect of AP303 on ECG parameters | Day 1-28
  Number of participants with abnormal heart rate

SECONDARY OUTCOMES:
Fasting glucose | Baseline, Days 6, 10, 14 and 28
  Change of fasting glucose
Fasting lipid profile | Baseline, Days 6, 10, 14 and 28
  Change of Triglyceride, HDL-C, LDL-C, Total cholesterol
Serum creatinine | Baseline, Days 6, 10, 14 and 28
  Change of serum creatinine
eGFR | Baseline, Days 6, 10, 14 and 28
  Change of estimated glomerular filtration rate

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zhang, Principal Investigator — Peking University First Hospital; Ying Gao, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No